CLINICAL TRIAL: NCT01708161
Title: A Phase Ib/II Study of the Combination of BYL719 Plus AMG 479 in Adult Patients With Selected Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719X2105J; 2012-001962-13 (EudraCT Number)
Record Dates: First submitted 2012-09-19; First posted 2012-10-16 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: PIK3CA Mutated Advanced Solid Tumors; PIK3CA Amplified Advanced Solid Tumors
Keywords: PIK3CA mutation; advanced solid tumor; breast cancer; ovarian cancer; cancers with a mass; bulky tumor; nodule; lump; advanced cancer; advanced solid malignancies
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Alpelisib; ganitumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BYL719 + AMG 479 (Experimental): For: Dose escalation phase/Phase II Expansion Phase. Cohorts of 3-6 patients were to be enrolled sequentially until an MTD or a recommended Phase II dose were defined. All patients were to receive the combination treatment. Sequential cohorts may receive different doses of the combination. In the Phase II expansion, all patients were to receive the same combination treatment.
  Interventions: Drug: BYL719; Drug: AMG 479

INTERVENTIONS:
Drug: BYL719 — BYL719 is a small molecule inhibiting PI3-Kinase.
  Other Names: ALPELISIB
Drug: AMG 479 — AMG 479 is a monoclonal antibody directed against IGF1-R.
  Other Names: ganitumab

SUMMARY:
This was a multi-center, open-label, phase Ib/II study. The aim of the phase Ib part was to estimate the MTD(s) and/or identify the recommended phase II dose(s) (RP2Ds) for the combination of BYL719 and AMG 479 (ganitumab), followed by the phase II part to assess the clinical efficacy and to further assess the safety of the combination in selected patient populations. Patients were to be treated until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. All patients were to be followed up. At a minimum, patients must have completed the safety follow-up assessments 30 days after the last dose of the study treatment.

DETAILED DESCRIPTION:
This was a multi-center, open-label, phase Ib/II study. The aim of the phase Ib part was to estimate the MTD(s) and/or identify the recommended phase II dose(s) (RP2Ds) for the combination of BYL719 and AMG 479 (ganitumab), followed by the phase II part to assess the clinical efficacy and to further assess the safety of the combination in selected patient populations. The dose escalation part of the study were to be guided by a Bayesian Logistic Regression Model (BLRM).

Once MTD/RP2D had been determined, patients were to be enrolled in two Phase II arms. Patients with PIK3CA mutated or amplified hormone receptor positive breast carcinoma were to be enrolled in Arm 1; patients with PIK3CA mutated or amplified ovarian carcinoma were to be enrolled in Arm 2. Patients were to be treated until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurred first. All patients were to be followed up. At a minimum, patients must have completed the safety follow-up assessments 30 days after the last dose of the study treatment.

ELIGIBILITY:
Key inclusion criteria:

* Written informed consent.
* Patients aged ≥ 18 years (male or female).
* Patients with the following histologically/cytologically-confirmed advanced solid tumors with documented somatic PIK3CA mutations or amplifications in tumor tissue:
* Hormone receptor positive breast carcinoma
* Ovarian carcinoma
* Other tumors upon agreement with sponsor
* Adequate organ function
* Negative serum pregnancy test

Key exclusion criteria:

* Patients with known history of severe infusion reactions to monoclonal antibodies.
* Patients with primary CNS tumor or CNS tumor involvement.
* History of thromboembolic event requiring full-dose anti-coagulation therapy any time prior to enrollment.
* Clinically significant cardiac disease.
* History of another malignancy within last 2 years.
* Pregnant or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-11-27 (Actual); Primary Completion 2014-12-26 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (4):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Nashville, Tennessee
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with selected advanced solid tumors who had relapsed or progressed on standard therapy were treated in BYL719X2105J study with a combination of alpelisib and ganitumab. Phase I of the trial was by dose combination of the treatment. Phase II was by patients.
Groups:
- BYL 200mg + AMG 12mg/kg; BYL 300mg + AMG 12mg/kg; BYL 350mg + AMG 12mg/kg: BYL719 (alpelisib) and AMG 479 (ganitumab) regimen in patients with PIK3CA mutated or amplified solid tumors
- HR+BC - Phase II: Patients with PIK3CA mutated or amplified hormone receptor (HR) positive breast carcinoma (BC) were treated with alpelisib 300 mg once daily and ganitumab 12 mg/kg.
- Ovarian - Phase II: Patients with PIK3CA mutated or amplified ovarian cancer were treated with alpelisib 300 mg once daily and ganitumab 12 mg/kg
- Non-HR+BC/Ovarian - Phase II: Patients with other than Breast and Ovarian cancer treated in the phase II part
Period: Overall Study
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg | HR+BC - Phase II | Ovarian - Phase II | Non-HR+BC/Ovarian - Phase II
Started | 4 | 10 | 10 | 16 | 6 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 10 | 10 | 16 | 6 | 1
Not completed — Adverse Event | 1 | 3 | 4 | 2 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Administrative problems | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Disease progression | 3 | 5 | 5 | 13 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg | HR+BC - Phase II | Ovarian - Phase II | Non-HR+BC/Ovarian - Phase II | Total
Number analyzed (Participants) | 4 | 10 | 10 | 16 | 6 | 1 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Full analysis set
  years | 50.5 (3.11) | 57.5 (15.55) | 63.7 (7.83) | 51.3 (8.04) | 59.7 (6.53) | 56.0 (0) | 56.3 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    Female | 4 | 7 | 7 | 15 | 6 | 1 | 40
    Male | 0 | 3 | 3 | 1 | 0 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 8 | 10 | 14 | 5 | 1 | 40
  Asian | 2 | 2 | 0 | 2 | 0 | 0 | 6
  Native American | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs) - Phase Ib
Description: Phase lb only
Time Frame: 28 days
Population: Dose determining set (DDS): DDS includes all patients from the safety set who either met the minimum treatment exposure and safety evaluation requirements without experiencing DLT within Cycle 1 or experienced a DLT at any time during Cycle 1.
Measure: Number; unit: Participants
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 3 | 8 | 9
Participants
  Drug hypersensitivity | 0 | 0 | 1
  Hyperglycemia | 0 | 0 | 1
  Rash maculopapular | 0 | 1 | 0
  Urticaria | 0 | 1 | 0

2. Primary Outcome: Percentage of Patients With Overall Response Rate (RECIST) Based on Investigator Radiology Assessment for HR Positive Breast and Ovarian Cancer - Phase II
Description: The antitumor activity of alpelisib in combination with ganitumab in patients with PIK3CA mutated or amplified hormone receptor positive (HR+) breast (arm 1) or ovarian (arm 2) cancer.
  Overall response rate is defined as the proportion of patients who have a best overall response of complete response or partial response assessed per RECIST 1.1.
Time Frame: Approximately 1 year (since initiation of Phase II, Dec 2013, till Primary CSR cut off 06Jan2015)
Population: Full analysis set (FAS). The full analysis set (FAS) includes all patients who received at least one full or partial dose of alpelisib or ganitumab. Patients were analyzed according to the planned treatment combination.
Measure: Number (95% Confidence Interval); unit: Percentages of participants
Groups:
- All Patients - Phase: The total column "All patients" includes a patient with non-HR+BC and non-Ovarian cancer treated in the Phase II part.
Arm/Group | HR+BC - Phase II | Ovarian - Phase II | All Patients - Phase
Number analyzed (Participants) | 16 | 6 | 23
Percentages of participants | 12.5 [1.6 to 38.3] | 16.7 [0.4 to 64.1] | 13.0 [2.8 to 33.6]

3. Secondary Outcome: Number of Patients With Best Overall Response (RECIST) Based on Investigator Radiology Assessment - Phase Ib
Description: The anti-tumor activity of alpelisib and ganitumab in combination as per RECIST 1.1
Time Frame: Approximately 1 year (since FPFV 27Nov2012, till MTD declaration 26Nov2013)
Population: Full Analysis set
Measure: Number; unit: Participants
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 10 | 10
Participants
  Complete response (CR) | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 3
  Stable disease (PD) | 1 | 3 | 2
  Progressive disease (PD) | 3 | 3 | 3
  Unknown | 0 | 4 | 2

4. Secondary Outcome: Percentage of Patients With Disease Control Rate (RECIST) Based on Investigator Radiology Assessment - Phase Ib
Description: The anti-tumor activity of alpelisib and ganitumab in combination as per RECIST 1.1
Time Frame: Approximately 1 year (since FPFV 27Nov2012, till MTD declaration 26Nov2013)
Population: Full Analysis set
Measure: Number (95% Confidence Interval); unit: Percentages of participants
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 33 | 10
Percentages of participants | 25.0 [0.6 to 80.6] | 9.1 [6.7 to 65.2] | 50.0 [18.7 to 81.3]

5. Secondary Outcome: Percentage of Patients With Disease Control Rate (RECIST) Based on Investigator Radiology Assessment for HR Positive Breast and Ovarian Cancer - Phase II
Description: the antitumor activity of alpelisib in combination with ganitumab in patients with PIK3CA mutated or amplified hormone receptor positive (HR+) breast (arm 1) or ovarian (arm 2) cancer.
  Phase II only, Cycle 1 Day 1 through Cycle 6 Day 28; assessed at baseline and every 8 weeks thereafter
Time Frame: Approximately 1 year (since initiation of Phase II, Dec 2013, till Primary CSR cut off 06Jan2015)
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentages of participants
Groups:
- All Patients - Phase II: The total column "All patients" includes a patient with non-HR+BC and non-Ovarian cancer treated in the Phase II part.
Arm/Group | HR+BC - Phase II | Ovarian - Phase II | All Patients - Phase II
Number analyzed (Participants) | 16 | 6 | 23
Percentages of participants | 43.8 [19.8 to 70.1] | 50.0 [11.8 to 88.2] | 47.8 [26.8 to 69.4]

6. Secondary Outcome: Cmax of BYL - Phase Ib
Description: Serum concentration for BYL719 (alpelisib)
  1 cycle - 28 days of treatment
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15
Population: Pharmacokinetic analysis set (PAS). The PAS included all patients who had at least one blood sample providing evaluable PK data. Patients were analyzed according to the dose level they actually received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 10 | 10
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 9 | 10
  Cycle 1 Day 1 | 2070 (1040) | 2620 (1260) | 2640 (888)
  Cycle 1 day 15: number analyzed (Participants) | 3 | 6 | 6
  Cycle 1 day 15 | 3080 (1750) | 2880 (910) | 2600 (1040)

7. Secondary Outcome: Area Under Curve (AUC) 0-24 Hour of BYL - Phase Ib
Description: Area under curve for BYL719 (alpelisib)
  1 cycle - 28 days of treatment
Time Frame: Cycle 1 Day 1 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post-dose), Cycle 1 Day 15 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post-dose)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 10 | 10
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 9 | 10
  Cycle 1 Day 1 | 19900 (8700) | 23400 (10500) | 25200 (9200)
  Cycle 1 day 15: number analyzed (Participants) | 3 | 6 | 6
  Cycle 1 day 15 | 24000 (10700) | 29700 (9170) | 25200 (9160)

8. Secondary Outcome: Tmax and T Half of BYL - Phase Ib
Description: Tmax and half life of BYL719 (Alpelisib)
  1 cycle - 28 days of treatment
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 10 | 10
hr
  Tmax (Cycle 1 Day 1): number analyzed (Participants) | 4 | 9 | 10
  Tmax (Cycle 1 Day 1) | 2.78 [1.88 to 3.55] | 1.97 [0.63 to 3.00] | 2.36 [1.50 to 3.10]
  Tmax (Cycle 1 Day 15): number analyzed (Participants) | 3 | 6 | 6
  Tmax (Cycle 1 Day 15) | 1.57 [0.83 to 1.83] | 3.01 [2.07 to 4.00] | 2.02 [2.00 to 3.08]
  Thalf (Cycle 1 Day 1): number analyzed (Participants) | 4 | 8 | 10
  Thalf (Cycle 1 Day 1) | 7.78 [6.24 to 10.80] | 6.06 [5.26 to 13.70] | 6.86 [5.32 to 9.23]
  Thalf (Cycle 1 Day15): number analyzed (Participants) | 3 | 6 | 6
  Thalf (Cycle 1 Day15) | 6.89 [5.94 to 9.90] | 6.80 [5.82 to 8.81] | 6.83 [5.19 to 13.00]

9. Secondary Outcome: Cmax of AMG - Phase Ib
Description: Serum concentration for AMG 479 (ganitumab)
  1 cycle - 28 days of treatment
Time Frame: Cycle 1 Day 15
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 10 | 10
ng/mL | 192 (24) | 202 (43.3) | 232 (59.3)

10. Secondary Outcome: Area Under Curve (AUC) 0-336 Hour of AMG - Phase Ib
Description: Area under curve for AMG 479 (ganitumab)
  1 cycle - 28 days of treatment
Time Frame: Cycle 1 Day 15 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post-dose)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 10 | 10
hr*ng/mL | 22900 (3930) | 22500 (7040) | 25200 (8000)

11. Secondary Outcome: Tmax and T Half of AMG - Phase Ib
Description: Tmax and half life of AMG 479 (ganitumab)
  1 cycle - 28 days of treatment
Time Frame: Cycle 1 Day 15
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | BYL 200mg + AMG 12mg/kg | BYL 300mg + AMG 12mg/kg | BYL 350mg + AMG 12mg/kg
Number analyzed (Participants) | 4 | 10 | 10
hr
  Tmax: number analyzed (Participants) | 3 | 8 | 9
  Tmax | 21.20 [1.02 to 22.70] | 1.02 [1.00 to 23.10] | 1.07 [1.00 to 1.77]
  Thalf: number analyzed (Participants) | 2 | 7 | 9
  Thalf | 132 [117 to 148] | 117 [109 to 161] | 180 [98 to 283]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 4.5 years.
Description: One patients with a tumor type other than Breast and Ovarian treated in the phase II part not represented.
Groups:
- BYL 200mg + AMG 12 mg/kg; BYL 300mg + AMG 12 mg/kg; BYL 350mg + AMG 12 mg/kg: BYL719 (alpelisib) and AMG 479 (ganitumab) regimen in patients with PIK3CA mutated or amplified solid tumors
- HR + BC - Phase II: Patients with PIK3CA mutated or amplified hormone receptor (HR) positive breat carcinoma (BC) were treated with alpelisib 300 mg once daily and ganitumab 12 mg/kg
- Ovarian - Phase II: Patients with other than Breast and Ovarian cancer treated in the phase II
Arm/Group | BYL 200mg + AMG 12 mg/kg | BYL 300mg + AMG 12 mg/kg | BYL 350mg + AMG 12 mg/kg | HR + BC - Phase II | Ovarian - Phase II
All-Cause Mortality (participants affected / at risk) | 4/4 | 8/10 | 8/10 | 13/16 | 5/6
Serious Adverse Events (participants affected / at risk) | 1/4 | 5/10 | 5/10 | 9/16 | 5/6
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 10/10 | 16/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYL 200mg + AMG 12 mg/kg (N=4) | BYL 300mg + AMG 12 mg/kg (N=10) | BYL 350mg + AMG 12 mg/kg (N=10) | HR + BC - Phase II (N=16) | Ovarian - Phase II (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BYL 200mg + AMG 12 mg/kg (N=4) | BYL 300mg + AMG 12 mg/kg (N=10) | BYL 350mg + AMG 12 mg/kg (N=10) | HR + BC - Phase II (N=16) | Ovarian - Phase II (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 2
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 2 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 7 | 10 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 3 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival erosion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 9 | 5 | 7 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 3 | 5 | 6 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 6 | 4 | 4 | 3
Asthenia (General disorders) | 0 | 2 | 2 | 3 | 3
Axillary pain (General disorders) | 0 | 0 | 0 | 2 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 2 | 3 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 6 | 8 | 7 | 2
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 0 | 1 | 0
Instillation site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 3 | 1
Oedema peripheral (General disorders) | 0 | 2 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 4 | 1
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasal herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 1 | 2
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 3 | 2 | 0 | 2
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 5 | 9 | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 6 | 8 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 5 | 4 | 4 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 7 | 9 | 9 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 5 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 3 | 2 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 4 | 4 | 3 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 5 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 2 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 4 | 2 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 6 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 5 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the competitive landscape for anticancer therapies in ovarian and breast cancer and given the limited clinical activity observed with the study combination treatment, Novartis decided in 2014 to halt the recruitment in the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.